CLINICAL TRIAL: NCT06070116
Title: Safety and Efficacy of Novel Combination Regimens for Treatment of Onchocerciasis
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Public Health Institute of Liberia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202307136
Record Dates: First submitted 2023-09-14; First posted 2023-10-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Onchocercal Subcutaneous Nodule; Onchocerciasis; Onchocerciasis, Ocular; Onchocerca Infection; Tropical Disease
MeSH Terms: conditions — Onchocerciasis; Onchocerciasis, Ocular | interventions — Albendazole; Ivermectin; Diethylcarbamazine; moxidectin

STUDY DESIGN:
Intervention Model Description: IVM + ALB (IA) - Dose of oral IVM (150 µg/kg) plus ALB (400 mg)
  Mox + ALB (MoxA) - Dose of oral Mox (8mg tablets) plus ALB (400mg)
  IVM + DEC + ALB (IDA) - Dose of oral IVM (150 µg/kg), DEC (6 mg/kg) and ALB (400 mg)
  MOX + DEC + IVM (MoxDA) - Dose of oral Mox (8 mg), DEC (6 mg/kg) and ALB (400 mg)
Masking Description: While this is an open label study and there is no placebo treatment group, all efforts will be made to ensure that that medical/technical staff assessing skin Mf, adverse events (AEs) and ophthalmological findings will be unaware of initial baseline skin and ocular Mf findings and treatment arm as best as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Ivermectin + Albendazole (IA) (Active Comparator): Dose of oral Ivermectin (150 µg/kg) plus Albendazole (400 mg)
  Interventions: Drug: Ivermectin w/ Albendazole
- Ivermectin + Diethylcarbamazine + Albendazole (IDA) (Experimental): Dose of oral Ivermectin (150 µg/kg), Diethylcarbamazine (6 mg/kg) and Albendazole (400 mg)
  Interventions: Drug: Ivermectin + Diethylcarbamazine + Albendazole
- Moxidectin + Albendazole (MoxA) (Experimental): Dose of oral Moxidectin (8mg) plus Albendazole (400 mg)
  Interventions: Drug: Moxidectin + Albendazole
- Moxidectin+ Diethylcarbamazine + Albendazole (MoxDA) (Experimental): Dose of oral Moxidectin (8mg), Diethylcarbamazine (6 mg/kg) and Albendazole (400 mg)
  Interventions: Drug: Moxidectin + Diethylcarbamazine + Albendazole

INTERVENTIONS:
Drug: Ivermectin w/ Albendazole — Participants will be given a dose of oral Ivermectin (IVM) (150 µg/kg) plus Albendazole (ALB) (400 mg)
  Other Names: IA
  Arms: Ivermectin + Albendazole (IA)
Drug: Ivermectin + Diethylcarbamazine + Albendazole — Participants will be given a dose of oral Ivermectin (IVM) (150 µg/kg), Diethylcarbamazine (DEC) (6 mg/kg) and Albendazole (ALB) (400 mg)
  Other Names: IDA
  Arms: Ivermectin + Diethylcarbamazine + Albendazole (IDA)
Drug: Moxidectin + Albendazole — Participants will be given a dose of oral Moxidectin (Mox) (8 mg) plus Albendazole (ALB) (400 mg)
  Other Names: MoxA
  Arms: Moxidectin + Albendazole (MoxA)
Drug: Moxidectin + Diethylcarbamazine + Albendazole — Participants will be given a dose of oral Moxidectin (Mox) (8 mg), Diethylcarbamazine (DEC) (6 mg/kg) and Albendazole (ALB) (400 mg)
  Other Names: MoxDA
  Arms: Moxidectin+ Diethylcarbamazine + Albendazole (MoxDA)

SUMMARY:
This study will investigate the safety and effectiveness of combination regimens in persons with onchocerciasis when it is administered after pre-treatment with ivermectin to clear or greatly reduce microfilariae from the skin and eyes.

DETAILED DESCRIPTION:
The open label, randomized clinical trial studies the safety and efficacy of combination regimens for the treatment of onchocerciasis. Around 300 participants from Bong Mines, Liberia will be randomly assigned to one of four treatment groups after receiving Ivermectin pre-treatment: Ivermectin plus Albendazole (IA0, Ivermectin plus DEC plus Albendazole (IDA), Moxidectin plus albendazole (MoxA), or Moxidectin plus DEC plus Albendazole (MoxDA). Participants will be treated at baseline and 6 months after initial treatment.

Safety will be measured through extensive adverse event monitoring from baseline to 6 months.

Efficacy of the treatment will be measured at 24 months after the initial treatment by the proportion of all adult female worms that are fertile in the Onchocerca nodules and the percentage of participants without microfilaremia at 6, 18, and 24 months after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women, 18 years to 75 years old
* Participants must have at least 1 palpable subcutaneous nodule (onchocercoma)
* Participants with mean skin Mf counts ≥ 1 Mf/mg at the time of enrollment (prior to pretreatment)

Exclusion Criteria:

* History of treatment with IVM or Mox less than six months prior to pretreatment with IVM.
* Treatment with IVM or Mox outside of the study after the pre-treatment clearing dose before treatment with one of the four study treatments.
* Pregnant or breastfeeding mothers.
* Severe ocular disease at baseline (assessed just prior to the first study treatment, approximately 6-12 months after IVM pretreatment). Briefly, these conditions include severe uveitis, severe glaucoma, severe keratitis, and/or cataracts that interfere with visualization of the posterior segment of the eye. Details regarding ocular exclusion criteria are provided below. Individuals who are excluded with significant ocular disease will be referred for appropriate All ocular disease exclusion criteria apply to either eye. That is to say, participants will be excluded if any of the ocular exclusion criteria listed below are met for either eye. These exclusions are needed to reduce the risk of study treatments worsening severe pre-existing ocular disease. They also are needed to ensure that study staff will be able to adequately evaluate the posterior segment before and after treatment.

  1. Any cataract that prevents clear visualization of fundus or imaging by OCT.
  2. Severe retinal nerve fiber layer thinning of the optic nerve in the superior and inferior quadrant analysis by OCT with a corresponding visual field defect in the superior and inferior hemifield, and/or visual field loss within 5 degrees of fixation in at least one hemifield. Note: If OCT is not available, the following exclusion criteria will apply: vertical cup/disc ratio by fundoscopy greater than or equal to 0.80 with a corresponding visual field defect in the superior and inferior hemifield, and/or visual field loss within 5 degrees of fixation in at least one hemifield.
  3. Intraocular pressure (IOP) greater than or equal to 25 by Goldmann tonometry.
  4. Retinal detachment or retinal break.
  5. Acute ocular infection (i.e., viral conjunctivitis, corneal ulcer, endophthalmitis).
  6. Optic atrophy with a reproducible visual field defect detected by confrontation visual field testing.
  7. Exam consistent with Herpes simplex virus eye infection.
  8. Homonymous hemianopsia, quadrantopsia, bitemporal hemianopsia, or central scotoma related to cerebral vascular disease by Automated Visual field testing and confrontation visual field testing.
  9. Acute angle closure glaucoma.
  10. Gonioscopy grade 0 (slit) limiting ability to safely dilate participant.
  11. Severe tremor, blepharospasm, or other voluntary or involuntary motor condition that limits careful slit lamp examinations, OCT, gonioscopy, IOP measurement, fundus photography, and automated perimetry.
  12. Cognitive impairment that limits participant's ability to understand and perform a Visual Acuity Test with a Tumbling E chart, confrontation visual field, slit lamp exam, or any other ocular exam component.
  13. Optic nerve edema.
  14. Active retinopathy or retinitis not attributable to onchocercal disease.
  15. A history of uveitis not associated with onchocerciasis.
  16. Any pre-existing chorioretinal scar or retinal degeneration and other significant retinal pathologies (foveomacular schisis, dystrophies, arterial macroaneurysms etc) involving the macula.
  17. Severe ocular pain that the participant rates as 9 or 10 out of 10.
  18. Best corrected or pinhole visual acuity worse than 6/60 (20/200).
  19. Age-related macular degeneration (AMD).
  20. >5 motile Mf in the anterior chamber in either eye at the time of secondary screening (6 months after pre-treatment with IVM).*
  21. The presence of one or more Mf in the posterior segment of the eye (detected by any opthalmological test performed) at the time of treatment (at least six months after pre-treatment with IVM). *Note regarding exclusion criteria t and u: The cut-off of 5 Mf in either anterior chamber was suggested by external reviewers of our proposal to the Gates Foundation. These were experts in onchocerciasis selected by the Foundation. The reviews were anonymous, so we do not know their names. They also suggested that we exclude persons with any Mf in the posterior segment of the eye, and we have added that exclusion criterion to the protocol.
* Significant comorbidities such as renal insufficiency (creatinine > 2 times the upper limit of normal), liver disease (jaundice or either AST or ALT greater than 2.5 times the upper limit of normal), or any other acute or chronic illness identified by study clinicians and investigators that interferes with the participant's ability to go to school or work or perform routine household chores.
* Prior allergic or hypersensitivity reactions or intolerance to IVM, Mox, ALB, or DEC.
* Evidence of severe or systemic comorbidities (aside from features of onchocerciasis), as judged by a study physician. Persons with baseline medical conditions that correspond to adverse event severity scores of grade 3 or higher will also be excluded.
* Evidence of urinary tract infection as indicated by 3+ nitrites by dipstick (individuals with 1+ or 2+ nitrites will not be excluded) or underlying chronic kidney disease as indicated by 3+ protein or 3+ blood by dipstick. Persons with urinary tract infections can be enrolled after their infections are treated and cured.
* Hgb <7 gm/dL; any such individuals will be referred to a local health center for evaluation and treatment).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Rates and types of severe or serious adverse events within 6 months following Ivermectin treatments | Baseline to 6 months
  Rates and types of severe or serious adverse events (grade 3 or higher) occurring within 6 months following combination treatment with DEC, ivermectin, and albendazole ("IDA") vs. the comparator regimen of ivermectin plus albendazole ("IA").
Rates and types of severe or serious adverse events within 6 months following Moxidectin treatments | Baseline to 6 months
  Rates and types of severe or serious adverse events (grade 3 or higher) occurring within 6 months following combination treatment with DEC, moxidectin, and albendazole ("MoxDA") vs. the comparator regimen of moxidectin plus albendazole ("MoxA").
Proportion of all adult female worms that are fertile 24 months after first treatment | 24 months
  Proportion of all adult female worms in nodules that are fertile (i.e. with morulae or later developmental stages in the uterus) 24 months after the first treatment dose. The primary objective efficacy analysis will be restricted to comparisons between IA vs IDA and between MoxA vs. MoxDA, respectively.

SECONDARY OUTCOMES:
Rates of adverse events grade 3 or higher by Ivermectin treatment group, that occur within 7 days of treatment | Baseline to 7 days after first treatment.
  Rates of adverse events grade 3 or higher by treatment group, that occur within 7 days of treatment. Comparison is made between IA vs IDA.
Rates of adverse events grade 3 or higher by Moxidectin treatment group, that occur within 7 days of treatment | Baseline to 7 days after first treatment.
  Rates of adverse events grade 3 or higher by treatment group, that occur within 7 days of treatment. Comparison is made between MoxA vs MoxDA.
Rates of adverse events grade 3 or higher in participants with ocular MF in Ivermectin treatment groups. | Baseline to 7 days after first treatment.
  Rates of adverse events grade 3 or higher that occur within 7 days of treatment in participants with detectable intraocular microfilariae just before the study treatment.
Rates of adverse events grade 3 or higher in participants with ocular MF in Moxidectin treatment groups. | Baseline to 7 days after first treatment.
  Rates of adverse events grade 3 or higher that occur within 7 days of treatment in participants with detectable intraocular microfilariae just before the study treatment.
Rates of ocular adverse events (any grade) by Ivermectin treatment group | Baseline to 7 days after first treatment.
  To compare rates of ocular adverse events (any grade) by treatment group that occur within 7 days of treatment. Comparison is between IA vs IDA.
Rates of ocular adverse events (any grade) by Moxidectin treatment groups | Baseline to 7 days after first treatment.
  To compare rates of ocular adverse events (any grade) by treatment group that occur within 7 days of treatment. Comparison is between MoxA vs MoxDA.
Percentage of adult female worms in nodules that are alive | 24 Months
  Percentage of adult female worms in nodules that are alive 24 months after the first round of study treatment.
Percentage of nodules with microfilaria in tissue | 24 Months
  The percentage of nodules with microfilariae in nodule tissue (outside of worms)
Percentage of nodules that do not contain living adult worms | 24 Months
  The percentage of nodules that do not contain any living adult female worms
Percentage of participants without microfiladermia after the first study treatment. | 6, 18, and 24 Months
  Percentage of participants without microfiladermia at 6, 18 and 24 months after the first study treatment.
Percentage of participants with recurrence of microfilariae in the skin across treatment groups | 18 and 24 Months
  Percentage of participants with recurrence of microfilariae in the skin at 18 and 24 months after the first study treatment (among persons who had complete Mf clearance 6 months after the first study treatment).
Microfilariae density in the skin across treatment groups | 6, 8, and 24 Months
  Mf density in the skin at 6, 18, and 24 months after the first study treatment.
Percentage of nodules with fully or partially calcified worms | 24 Months
  Percentage of nodules with fully or partially calcified worms 24 months after the first round of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Fischer, PhD, Principal Investigator — Washington University School of Medicine; Patrick Kpanyen, PhD, Principal Investigator — National Public Health Institute of Liberia; Gary Weil, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Bong County Hospital, Bong Town, Bong County, Liberia

IPD SHARING:
Plan to Share IPD: Yes
Datasets used for published results will be shared publicly through the Washington University School of Medicine Becker Library so that the broader scientific community can access it. Only de-identified data will be shared publicly.
Supporting Information: Study Protocol, SAP
Time Frame: Dataset will be shared through Washington University School of Medicine Becker Library at the time of publication.

REFERENCES:
- [Background] Herricks JR, Hotez PJ, Wanga V, Coffeng LE, Haagsma JA, Basanez MG, Buckle G, Budke CM, Carabin H, Fevre EM, Furst T, Halasa YA, King CH, Murdoch ME, Ramaiah KD, Shepard DS, Stolk WA, Undurraga EA, Stanaway JD, Naghavi M, Murray CJL. The global burden of disease study 2013: What does it mean for the NTDs? PLoS Negl Trop Dis. 2017 Aug 3;11(8):e0005424. doi: 10.1371/journal.pntd.0005424. eCollection 2017 Aug. No abstract available. PMID 28771480
- [Background] Taylor MJ, Awadzi K, Basanez MG, Biritwum N, Boakye D, Boatin B, Bockarie M, Churcher TS, Debrah A, Edwards G, Hoerauf A, Mand S, Matthews G, Osei-Atweneboana M, Prichard RK, Wanji S, Adjei O. Onchocerciasis Control: Vision for the Future from a Ghanian perspective. Parasit Vectors. 2009 Jan 21;2(1):7. doi: 10.1186/1756-3305-2-7. PMID 19154624
- [Background] Zimmerman PA, Dadzie KY, De Sole G, Remme J, Alley ES, Unnasch TR. Onchocerca volvulus DNA probe classification correlates with epidemiologic patterns of blindness. J Infect Dis. 1992 May;165(5):964-8. doi: 10.1093/infdis/165.5.964. PMID 1569351
- [Background] Fischer P, Kipp W, Bamuhiga J, Binta-Kahwa J, Kiefer A, Buttner DW. Parasitological and clinical characterization of Simulium neavei-transmitted onchocerciasis in western Uganda. Trop Med Parasitol. 1993 Dec;44(4):311-21. PMID 8134773
- [Background] Dadzie KY, Bird AC, Awadzi K, Schulz-Key H, Gilles HM, Aziz MA. Ocular findings in a double-blind study of ivermectin versus diethylcarbamazine versus placebo in the treatment of onchocerciasis. Br J Ophthalmol. 1987 Feb;71(2):78-85. doi: 10.1136/bjo.71.2.78. PMID 3548811
- [Background] Taylor HR. Onchocerciasis. Int Ophthalmol. 1990 May;14(3):189-94. doi: 10.1007/BF00158317. PMID 2188920
- [Background] Bird AC, el-Sheikh H, Anderson J, Fuglsang H. Changes in visual function and in the posterior segment of the eye during treatment of onchocerciasis with diethylcarbamazine citrate. Br J Ophthalmol. 1980 Mar;64(3):191-200. doi: 10.1136/bjo.64.3.191. PMID 7387952
- [Background] Duke BO. Human onchocerciasis--an overview of the disease. Acta Leiden. 1990;59(1-2):9-24. PMID 2198761
- [Background] Braun G, McKechnie NM, Connor V, Gilbert CE, Engelbrecht F, Whitworth JA, Taylor DW. Immunological crossreactivity between a cloned antigen of Onchocerca volvulus and a component of the retinal pigment epithelium. J Exp Med. 1991 Jul 1;174(1):169-77. doi: 10.1084/jem.174.1.169. PMID 2056276
- [Background] Chandrashekar R, Curtis KC, Weil GJ. Molecular characterization of a parasite antigen in sera from onchocerciasis patients that is immunologically cross-reactive with human keratin. J Infect Dis. 1995 Jun;171(6):1586-92. doi: 10.1093/infdis/171.6.1586. PMID 7539474
- [Background] Chandrashekar R, Ogunrinade AF, Alvarez RM, Kale OO, Weil GJ. Circulating immune complex-associated parasite antigens in human onchocerciasis. J Infect Dis. 1990 Nov;162(5):1159-64. doi: 10.1093/infdis/162.5.1159. PMID 2230240
- [Background] Johnson TP, Tyagi R, Lee PR, Lee MH, Johnson KR, Kowalak J, Elkahloun A, Medynets M, Hategan A, Kubofcik J, Sejvar J, Ratto J, Bunga S, Makumbi I, Aceng JR, Nutman TB, Dowell SF, Nath A. Nodding syndrome may be an autoimmune reaction to the parasitic worm Onchocerca volvulus. Sci Transl Med. 2017 Feb 15;9(377):eaaf6953. doi: 10.1126/scitranslmed.aaf6953. PMID 28202777
- [Background] Kawabata M, Izui S, Anan S, Kondo S, Fukumoto S, Flores GZ, Kobayakawa T. Circulating immune complexes and their possible relevance to other immunological parameters in Guatemalan onchocerciasis. Int Arch Allergy Appl Immunol. 1983;72(2):128-33. doi: 10.1159/000234854. PMID 6874107
- [Background] Semba RD, Murphy RP, Newland HS, Awadzi K, Greene BM, Taylor HR. Longitudinal study of lesions of the posterior segment in onchocerciasis. Ophthalmology. 1990 Oct;97(10):1334-41. doi: 10.1016/s0161-6420(90)32413-2. PMID 2243684
- [Background] Banla M, Tchalim S, Karabou PK, Gantin RG, Agba AI, Kere-Banla A, Helling-Giese G, Heuschkel C, Schulz-Key H, Soboslay PT. Sustainable control of onchocerciasis: ocular pathology in onchocerciasis patients treated annually with ivermectin for 23 years: a cohort study. PLoS One. 2014 Jun 2;9(6):e98411. doi: 10.1371/journal.pone.0098411. eCollection 2014. PMID 24887413
- [Background] Diawara L, Traore MO, Badji A, Bissan Y, Doumbia K, Goita SF, Konate L, Mounkoro K, Sarr MD, Seck AF, Toe L, Touree S, Remme JH. Feasibility of onchocerciasis elimination with ivermectin treatment in endemic foci in Africa: first evidence from studies in Mali and Senegal. PLoS Negl Trop Dis. 2009 Jul 21;3(7):e497. doi: 10.1371/journal.pntd.0000497. PMID 19621091
- [Background] Rodriguez-Perez MA, Fernandez-Santos NA, Orozco-Algarra ME, Rodriguez-Atanacio JA, Dominguez-Vazquez A, Rodriguez-Morales KB, Real-Najarro O, Prado-Velasco FG, Cupp EW, Richards FO Jr, Hassan HK, Gonzalez-Roldan JF, Kuri-Morales PA, Unnasch TR. Elimination of Onchocerciasis from Mexico. PLoS Negl Trop Dis. 2015 Jul 10;9(7):e0003922. doi: 10.1371/journal.pntd.0003922. eCollection 2015. PMID 26161558
- [Background] Zarroug IM, Hashim K, ElMubark WA, Shumo ZA, Salih KA, ElNojomi NA, Awad HA, Aziz N, Katabarwa M, Hassan HK, Unnasch TR, Mackenzie CD, Richards F, Higazi TB. The First Confirmed Elimination of an Onchocerciasis Focus in Africa: Abu Hamed, Sudan. Am J Trop Med Hyg. 2016 Nov 2;95(5):1037-1040. doi: 10.4269/ajtmh.16-0274. Epub 2016 Jun 27. PMID 27352878
- [Background] Katabarwa MN, Eyamba A, Nwane P, Enyong P, Kamgno J, Kuete T, Yaya S, Aboutou R, Mukenge L, Kafando C, Siaka C, Mkpouwoueiko S, Ngangue D, Biholong BD, Andze GO. Fifteen years of annual mass treatment of onchocerciasis with ivermectin have not interrupted transmission in the west region of cameroon. J Parasitol Res. 2013;2013:420928. doi: 10.1155/2013/420928. Epub 2013 Apr 17. PMID 23691275
- [Background] Evans DS, Unnasch TR, Richards FO. Onchocerciasis and lymphatic filariasis elimination in Africa: it's about time. Lancet. 2015 May 30;385(9983):2151-2. doi: 10.1016/S0140-6736(15)61022-4. No abstract available. PMID 26068266
- [Background] Fischer PU, King CL, Jacobson JA, Weil GJ. Potential Value of Triple Drug Therapy with Ivermectin, Diethylcarbamazine, and Albendazole (IDA) to Accelerate Elimination of Lymphatic Filariasis and Onchocerciasis in Africa. PLoS Negl Trop Dis. 2017 Jan 5;11(1):e0005163. doi: 10.1371/journal.pntd.0005163. eCollection 2017 Jan. No abstract available. PMID 28056015
- [Background] Taylor HR, George T. Microfilaria in the cornea in onchocerciasis. Trans R Soc Trop Med Hyg. 1987;81(1):148. doi: 10.1016/0035-9203(87)90308-7. No abstract available. PMID 3445302
- [Background] Greene BM, Taylor HR, Brown EJ, Humphrey RL, Lawley TJ. Ocular and systemic complications of diethylcarbamazine therapy for onchocerciasis: association with circulating immune complexes. J Infect Dis. 1983 May;147(5):890-7. doi: 10.1093/infdis/147.5.890. PMID 6842023
- [Background] Greene BM, Taylor HR, Cupp EW, Murphy RP, White AT, Aziz MA, Schulz-Key H, D'Anna SA, Newland HS, Goldschmidt LP, et al. Comparison of ivermectin and diethylcarbamazine in the treatment of onchocerciasis. N Engl J Med. 1985 Jul 18;313(3):133-8. doi: 10.1056/NEJM198507183130301. PMID 3892293
- [Background] Basanez MG, Pion SD, Boakes E, Filipe JA, Churcher TS, Boussinesq M. Effect of single-dose ivermectin on Onchocerca volvulus: a systematic review and meta-analysis. Lancet Infect Dis. 2008 May;8(5):310-22. doi: 10.1016/S1473-3099(08)70099-9. PMID 18471776
- [Background] Awadzi K, Opoku NO, Attah SK, Lazdins-Helds J, Kuesel AC. A randomized, single-ascending-dose, ivermectin-controlled, double-blind study of moxidectin in Onchocerca volvulus infection. PLoS Negl Trop Dis. 2014 Jun 26;8(6):e2953. doi: 10.1371/journal.pntd.0002953. eCollection 2014 Jun. PMID 24968000
- [Background] Taylor HR. Ivermectin treatment of ocular onchocerciasis. Acta Leiden. 1990;59(1-2):201-6. PMID 2198751
- [Background] Taylor HR, Semba RD, Newland HS, Keyvan-Larijani E, White A, Dukuly Z, Greene BM. Ivermectin treatment of patients with severe ocular onchocerciasis. Am J Trop Med Hyg. 1989 May;40(5):494-500. doi: 10.4269/ajtmh.1989.40.494. PMID 2658637
- [Background] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704
- [Background] Awadzi K, Gilles HM. Diethylcarbamazine in the treatment of patients with onchocerciasis. Br J Clin Pharmacol. 1992 Oct;34(4):281-8. doi: 10.1111/j.1365-2125.1992.tb05632.x. No abstract available. PMID 1457260
- [Background] Opoku NO, Bakajika DK, Kanza EM, Howard H, Mambandu GL, Nyathirombo A, Nigo MM, Kasonia K, Masembe SL, Mumbere M, Kataliko K, Larbelee JP, Kpawor M, Bolay KM, Bolay F, Asare S, Attah SK, Olipoh G, Vaillant M, Halleux CM, Kuesel AC. Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial. Lancet. 2018 Oct 6;392(10154):1207-1216. doi: 10.1016/S0140-6736(17)32844-1. Epub 2018 Jan 18. PMID 29361335
- [Background] Opoku NO, Doe F, Dubben B, Fetcho N, Fischer K, Fischer PU, Gordor S, Goss CW, Gyasi ME, Hoerauf A, Hong AR, Kanza E, King CL, Laryea R, Lew D, Seidu MA, Weil GJ. A randomized, open-label study of the tolerability and efficacy of one or three daily doses of ivermectin plus diethylcarbamazine and albendazole (IDA) versus one dose of ivermectin plus albendazole (IA) for treatment of onchocerciasis. PLoS Negl Trop Dis. 2023 May 19;17(5):e0011365. doi: 10.1371/journal.pntd.0011365. eCollection 2023 May. PMID 37205721
- [Background] Wojtkowski M, Bajraszewski T, Gorczynska I, Targowski P, Kowalczyk A, Wasilewski W, Radzewicz C. Ophthalmic imaging by spectral optical coherence tomography. Am J Ophthalmol. 2004 Sep;138(3):412-9. doi: 10.1016/j.ajo.2004.04.049. PMID 15364223
- [Background] Jolodar A, Fischer P, Buttner DW, Miller DJ, Schmetz C, Brattig NW. Onchocerca volvulus: expression and immunolocalization of a nematode cathepsin D-like lysosomal aspartic protease. Exp Parasitol. 2004 Jul-Aug;107(3-4):145-56. doi: 10.1016/j.exppara.2004.06.006. PMID 15363940
- [Background] Lloyd MM, Gilbert R, Taha NT, Weil GJ, Meite A, Kouakou IM, Fischer PU. Conventional parasitology and DNA-based diagnostic methods for onchocerciasis elimination programmes. Acta Trop. 2015 Jun;146:114-8. doi: 10.1016/j.actatropica.2015.03.019. Epub 2015 Mar 25. PMID 25818324
- [Background] Edi C, Bjerum CM, Ouattara AF, Chhonker YS, Penali LK, Meite A, Koudou BG, Weil GJ, King CL, Murry DJ. Pharmacokinetics, safety, and efficacy of a single co-administered dose of diethylcarbamazine, albendazole and ivermectin in adults with and without Wuchereria bancrofti infection in Cote d'Ivoire. PLoS Negl Trop Dis. 2019 May 20;13(5):e0007325. doi: 10.1371/journal.pntd.0007325. eCollection 2019 May. PMID 31107869